CLINICAL TRIAL: NCT06127134
Title: Outcomes of Straight-line Flow Versus Angiosome-targeted Angioplasty in Treatment of Critical Lower Limb Ischemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Elsaid Hassan Bedeer, Principal Investigator, Kafrelsheikh University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MSKU 50-2-28
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Angioplasty; Critical Lower Limb Ischemia
Keywords: angioplasty; critical lower limb ischemia; chronic lower limb threatening ischemia; straight line; angiosome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Straight-line flow (Group A) (Active Comparator): treating less diseased arteries which is in line with distal run off the foot
  Interventions: Procedure: peripheral angioplasty for tibial vessels
- Angiosome-targeted (Group B) (Sham Comparator): treating specific angiosome through a targeted vessel which mainly supplies this angiosome
  Interventions: Procedure: peripheral angioplasty for tibial vessels

INTERVENTIONS:
Procedure: peripheral angioplasty for tibial vessels — repair tibials blood vessels throughout two concepts using angioplasty ballooning
  Other Names: endovascular arterial repair for critical lower limb ischemia

SUMMARY:
Peripheral arterial disease (PAD) affects more than 200 million people worldwide. Although over 50% are asymptomatic, it accounts for 4% of all amputations.

The ischemic limb must be revascularized to help wound healing, reduce the pain of ischemia and preserve the limb's function. So, surgical and percutaneous revascularization choices must be considered in CLI. Classically, CLI revascularization aims to provide at least one patent vessel that delivers in-line flow to the foot.

Today, the investigators live in a new era of angioplasty evolving and substituting open vascular surgery, so expanding research on endovascular strategy has been noticed.This confirms the profound impact of angioplasty in vascular surgery as one of the fastest-growing branches of medicine

Infrapopliteal artery occlusive disease (IPOD) is a significant cause of critical limb-threatening ischemia (CLTI). The worldwide prevalence of IPOD is between 4.5% and 29%, and most patients live in low-income countries.

The angiosomal concept was derived from plastic surgery for the skin flap. This concept delineates the human body into three-dimensional blocks of tissue from the skin to bone and also provides practical application of vascular anatomy for reconstructive surgery. An angiosome is an anatomic unit of tissue consisting of skin, subcutaneous, muscle, and bone fed by a source artery and drained by a specific vein.

According to the angiosomal concept, the foot is divided into six distinct angiosomes fed by source arteries, three from the posterior tibial, two from the peroneal, and one from the anterior tibial artery, with functional artery-to-artery connections among muscle, fascia, and skin. Numerous direct inter-arterial connections occur between the foot's main arteries, which provide alternative pathways of blood flow when disruption or compromise affects the arteries that directly feed the angiosome.

On the other hand, in patients with CLI, where only one vessel runoff can be established to the foot, direct flow into a patent pedal arch is essential to improve their clinical outcomes.

Conventional Endovascular therapy aims to the re-establishment of pulsatile straight-line flow to the lower limb. This results in relieving ischemic pain, healing ulcers, achieving limb salvage, improving quality of life, and potentially prolonging survival.

So it became essential to know the differential impact of both concepts on CLI revascularization.

DETAILED DESCRIPTION:
Introduction

Peripheral arterial disease (PAD) affects more than 200 million people worldwide. Although over 50% are asymptomatic, it accounts for 4% of all amputations.

The ischemic limb must be revascularized to help wound healing, reduce the pain of ischemia and preserve the limb's function. So, surgical and percutaneous revascularization choices must be considered in CLI. Classically, CLI revascularization aims to provide at least one patent vessel that delivers in-line flow to the foot.

Today, the investigators live in a new era of angioplasty evolving and substituting open vascular surgery, so expanding research on endovascular strategy has been noticed.This confirms the profound impact of angioplasty in vascular surgery as one of the fastest-growing branches of medicine

Infrapopliteal artery occlusive disease (IPOD) is a significant cause of critical limb-threatening ischemia (CLTI). The worldwide prevalence of IPOD is between 4.5% and 29%, and most patients live in low-income countries.

The angiosomal concept was derived from plastic surgery for the skin flap. This concept delineates the human body into three-dimensional blocks of tissue from the skin to bone and also provides practical application of vascular anatomy for reconstructive surgery. An angiosome is an anatomic unit of tissue consisting of skin, subcutaneous, muscle, and bone fed by a source artery and drained by a specific vein.

According to the angiosomal concept, the foot is divided into six distinct angiosomes fed by source arteries, three from the posterior tibial, two from the peroneal, and one from the anterior tibial artery, with functional artery-to-artery connections among muscle, fascia, and skin. Numerous direct inter-arterial connections occur between the foot's main arteries, which provide alternative pathways of blood flow when disruption or compromise affects the arteries that directly feed the angiosome.

On the other hand, in patients with CLI, where only one vessel runoff can be established to the foot, direct flow into a patent pedal arch is essential to improve their clinical outcomes.

Conventional Endovascular therapy aims to the re-establishment of pulsatile straight-line flow to the lower limb. This results in relieving ischemic pain, healing ulcers, achieving limb salvage, improving quality of life, and potentially prolonging survival.

So it became essential to know the differential impact of both concepts on CLI revascularization.

Aim of the work Comparing the efficiency of two percutaneous transluminal angioplasty techniques for Critical Lower Limb Ischemia revascularization, Straight-line flow (Group A) versus Angiosome-targeted (Group B).As regard short-term impact.

Patient and methods

1. Study Ethics the investigators will conduct this study after the approval of the I.R.B. (Institutional Review Board) of Kafrelsheikh University Hospital. All included procedures will be according to the Declaration of Helsinki. the investigators will also obtain the patients' informed consent to use their data in their research. All evaluation forms, reports, and other records that leave the site would not include unique personal data to maintain subject confidentiality.
2. Study design: a non-randomized clinical trial.
3. Time of study: The study will be conducted in 2023.
4. all patients will be submitted to the following preoperative evaluation : 1-History : 1. Personal data. 2. Risk factors: smoking, DM, hypertension, hypercholesterolemia. 3. Co-morbidity: previous stroke, angina, MI, and CKD. 4. Previous PAD interventions to one or both legs. 5. Previous amputations. 6. Previous coronary intervention (CABG, PCI) 2- Physical examination, including:

1. Assessment of functional status: independent stick walker, prosthesis, wheelchair, bed-bound 2. Recording of peripheral pulses 3. Measurement of ABPI or TBPI 4. Wound assessment (in those patients with tissue loss) 5. Assessment of ischaemic night/rest pain. 3-Investigations: A) Laboratory

1. Routine hematology (hemoglobin, white cell count, platelet count, HbA1c)
2. Routine biochemistry (creatinine, estimated GFR, ESR, CRP, RBS, cholesterol, HBA1c)
3. PT, PTT, INR
4. Lipid profile.

B)Imaging of their arteries by one or more of the following modalities:

1. Duplex ultrasound.
2. Computerized tomography angiography (CTA)
3. Magnetic resonance angiography (MRA)
4. Digital subtraction angiography (DUS)

(5) Patients with critical lower limb ischemia are going to be classified according to

• Modified TASC II classification 2016 (Trans-Atlantic Inter-society Consensus), which is a morphological classification

• Rutherford classification, which is the clinical classification

(6) Surgical procedure. Therapeutic intervention (angioplasty)

(7) Post-operative follow-up.

Follow-up of the patients will be at the first, third, and sixth months from the intervention date. Progress of limb conditions after the intervention will be observed which will be regarding :

* Diminution or absence of rest pain
* Healing of ulcers.
* limb salvage Assessed by Visual Analogue Scale (VAS)
* complications

  (8) Sampling technique:

The sample size of 100 patients classified into two groups

(9) Statistical analysis:

Analysis of data will be done using SPSS (statistical package for social science)

(10) Inclusion Criteria:

* Patient with documented symptomatic infragenicular chronic arterial disease with or without supra-genicular lesion
* Diabetic or not
* Rutherford grades 4, 5 and 6
* The patient is able and willing to comply with study follow-up requirements.

  (11) Exclusion Criteria:
* Contraindication for angioplasty
* unsuitable for angioplasty revascularization strategy
* claudication case
* tissue loss is considered to be primarily of venous etiology.
* Patient with full-thickness gangrene of the foot.
* Widespread infection of the lower limb needing amputation

  (12) Outcome Measures :
* Technical success as documented by angiography pre & post procedure with residual stenosis <30%
* Clinical success is improving at least one class in Rutherford classification in patients with chronic limb ischemia.
* Primary patency at six months follow-up.
* Successful target lesion revascularization.
* The absence of major adverse events is defined as unplanned major amputation of the index limb.
* Absence of non-managed complications

ELIGIBILITY:
Inclusion Criteria:

* Patient with documented symptomatic infragenicular chronic arterial disease with or without supra-genicular lesion
* Diabetic or not
* Rutherford grades 4, 5 and 6
* The patient is able and willing to comply with study follow-up requirements.

Exclusion Criteria:

* Contraindication for angioplasty
* unsuitable for angioplasty revascularization strategy
* claudication case
* tissue loss is considered to be primarily of venous etiology.
* Patient with full-thickness gangrene of the foot.
* Widespread infection of the lower limb needing amputation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Technical success | first 24 hours
  good distal flow and arterial pulsation which are documented by angiography pre & post procedure with residual stenosis <30%
Clinical success | first 6 month
  limb salvage and wound status improves at least one class in Rutherford classification in patients with critical limb ischemia.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Bedeer, MD, Principal Investigator — KFS university
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: Undecided